CLINICAL TRIAL: NCT07197489
Title: Prioritization of Patients With Suspected Acute Appendicitis Using the Appendistat Score (APS)
Brief Title: Prioritisation of Acute Appendicitis Using Appendistat Score
Acronym: APEX
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 206417
Record Dates: First submitted 2025-09-09; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Acute Appendicitis; Acute Appendicitis With Rupture
Keywords: Appendicitis; Appendistat score; Triage tool; risk stratification; complicated appendicitis; Emergency surgery
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Right iliac fossa pain: Post operative classification into: acute uncomplicated appendicitis; acute complicated appendicitis; and normal appendix

SUMMARY:
Introduction

Although non-operative management of acute appendicitis may be appropriate in selected cases, surgery remains the gold standard treatment. Prioritization of patients at risk of developing complicated appendicitis is essential for improving outcomes. The aim of this study was to assess the predictive value and clinical utility of the Appendistat (APS) scoring system as a triaging tool to prioritize patients with a high risk of developing complicated appendicitis.

Methods This was a chart review, cross-sectional observational diagnostic study, with a single-gate retrospective design, including 592 patients who underwent appendicectomy. Based on final histological diagnosis, patients were categorized as normal, acute uncomplicated appendicitis (AUA), or acute complicated appendicitis (ACA). The predictive value matrix of the APS score for identifying patients with a histological diagnosis of complicated appendicitis was calculated.

DETAILED DESCRIPTION:
Detailed Description

Introduction Although conservative treatment for acute appendicitis may be appropriate in selected patients, appendicectomy remains the gold standard treatment of choice for acute appendicitis, as advocated by clinical guidelines (1,2). The timing of surgery is critical for improving patient outcomes. Guidelines from the National Confidential Inquiry into Patient Outcome and Death (NCEPOD) in the UK recommend prompt surgical intervention within hours of presentation (NCEPOD Category 2) (3). Evidence suggests that delays beyond 24 hours are associated with considerable safety concerns (4,5). Specifically, postponing surgical treatment beyond this timeframe can increase the likelihood of appendiceal perforation, necrosis, gangrene, and postoperative complications (6). Westfall and Charles demonstrated that the relative risk of perforation increases by 9% for each day of delayed treatment (7). However, challenges in emergency theatre capacity across NHS trusts frequently result in delays exceeding 24 hours, placing patients at risk of progression from uncomplicated to complicated appendicitis. A triaging tool capable of predicting patients at high risk of perforation is therefore required to ensure prioritization for timely surgical intervention.

The Appendistat (APS) scoring system was developed to identify patients at risk of complicated appendicitis. The score employs a logistic regression analysis of objective variables, including age, sex, white cell count (WCC), C-reactive protein (CRP), and bilirubin, to identify patients likely to develop complicated appendicitis (8). The APS score can be readily calculated during the initial assessment of patients suspected of acute appendicitis and can be integrated into electronic patient record (EPR) systems without the need to include symptoms, signs, or imaging results.

The purpose of this study was to assess the predictive value and clinical utility of the APS score in identifying patients at risk of complicated appendicitis on admission to a busy surgical emergency unit (SEU) at John Radcliffe Hospital, Oxford.

Methods

Design and Patients This was a retrospective chart review, cross-sectional observational diagnostic study with a single-gate design. A total of 592 patients undergoing appendicectomy at John Radcliffe Hospital, Oxford, between April 2023 and April 2024 were included. Patients were identified retrospectively from the EPR (Cerner Millennium within BT Local Service Provider [LSP]). Approval was obtained from the Trust Clinical Governance Department (reference 9210). Data were anonymized by two clinicians (TPJ and GK) and analysed by the senior investigator (ME), who was blinded to patient identifiers.

Inclusion criteria were: patients aged ≥16 years with a conclusive histological report of the appendix.

Exclusion criteria were: elective appendicectomy, appendicectomy performed as part of another procedure (e.g., hysterectomy), or absence of definitive histopathology.

Data Collection Data extracted included demographics, preoperative WCC, CRP, bilirubin, imaging reports, time from admission to surgery, intraoperative findings, operative duration, postoperative hospital stay, and final histology.

Outcome Groups

Histological diagnosis was used as the reference standard. Three categories were defined by consultant pathologists:

* Normal appendix: no inflammation.
* Acute uncomplicated appendicitis (AUA): suppurative/phlegmonous with transmural inflammation, ulceration, thrombosis, or intramural pus.
* Acute complicated appendicitis (ACA): gangrenous, perforated, or transmural inflammation with intramural/extramural pus.

  1. Primary Outcome
* Title: Area under the ROC curve (AUC) of the Appendistat Score (APS) for predicting histologically confirmed complicated appendicitis.
* Description: Diagnostic accuracy of APS calculated using ROC and AUC analyses.
* Time Frame: At time of hospital admission (within 24 hours of presentation).
* Safety issue: No

  2. Secondary Outcome 1
* Title: Sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) of the Appendistat Score (APS) for detecting complicated appendicitis.
* Description: Diagnostic performance of APS compared with histology, expressed as sensitivity, specificity, PPV, and NPV at the defined cut-off point.
* Time Frame: At the time of hospital admission (within 24 hours of presentation).
* Safety issue: No

  3. Secondary Outcome 2
* Title: Mean Appendistat Score (APS) values in patients with acute uncomplicated vs. complicated appendicitis
* Description: Comparison of mean APS values between patients with histologically confirmed acute uncomplicated appendicitis and those with acute complicated appendicitis.
* Time Frame: At time of hospital admission (within 24 hours of presentation)
* Safety Issue: No

Statistical analysis

Data were analysed using the Statistical Package for the Social Sciences (SPSS) version 23 and GraphPad Prism version 10. Continuous variables were analysed with the t-test, and categorical variables with the chi-square test. Receiver operating characteristic (ROC) curve and area under the curve (AUC) analyses were used to establish the diagnostic accuracy and determine the cut-off point of the APS score for ACA. The score was calculated using WCC, CRP, and bilirubin values at first presentation. A p-value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 16-years and above, with a conclusive histological report were included.

Exclusion Criteria:

hysterectomy, and those without a conclusive pathology report were excluded

Ages: 16 Years to 95 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to the surgical assessment unit with acute right iliac fossa pain
Sampling Method: Probability Sample
Enrollment: 592 (Actual)
Dates: Start 2024-01-06 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2025-08-02 (Actual)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic (ROC) curve (AUC) of the Appendistat Score (APS) for predicting histologically confirmed complicated appendicitis | At time of hospital admission (within 24 hours of presentation)
  Diagnostic accuracy of APS assessed by calculating the AUC of the ROC curve for discriminating complicated appendicitis from

SECONDARY OUTCOMES:
Sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) of the Appendistat Score (APS) for detecting complicated appendicitis | At time of hospital admission (within 24 hours of presentation)
  Diagnostic performance of APS compared with histology, reported as sensitivity, specificity, PPV, and NPV at the defined cut-off value.
Mean Appendistat Score (APS) values in patients with histologically confirmed uncomplicated vs. complicated appendicitis | At time of hospital admission (within 24 hours of presentation)
  Comparison of mean APS values between patients with acute uncomplicated appendicitis and those with acute complicated appendicitis, based on histological diagnosis

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - University College London, London
  - Oxford University Hospitals NHS Trust, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lerea KM, Livingston JN. The different receptor species of liver have similar complex insulin binding properties. Biochem Biophys Res Commun. 1983 Aug 12;114(3):1042-7. doi: 10.1016/0006-291x(83)90667-8. PMID 6351858